CLINICAL TRIAL: NCT04724746
Title: Open Pilot Trial of an Integrated Intervention for Substance Use and Posttraumatic Stress Following Sexual Assault
Brief Title: Integrated Intervention Post-Sexual Assault
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Christine Hahn, Research Assistant Professor, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro0009631
Record Dates: First submitted 2021-01-21; First posted 2021-01-26 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Substance Use Disorders; Posttraumatic Stress Disorder; Sexual Assault
MeSH Terms: conditions — Substance-Related Disorders; Stress Disorders, Post-Traumatic | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Written Exposure and Cognitive Behavioral Therapy (Experimental): Participants receive 5 to 6, 60 minute, sessions of written exposure therapy for posttraumatic stress disorder combined with cognitive behavioral therapy for substance use disorder.
  Interventions: Behavioral: Written Exposure and Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Written Exposure and Cognitive Behavioral Therapy — Intervention involves writing details about a recent sexual assault and coping skills for substance use.

SUMMARY:
The primary objective of the proposed Stage IA/IB study is to establish feasibility of an integrated cognitive-behavioral intervention for reducing SUD and PTSD symptoms among women who experienced a sexual assault within the past six weeks. The intervention will be tested in an open label trial to make final modifications to evaluate feasibility, acceptability, and preliminary efficacy of the five to six week integrated intervention with standardized repeated measures during a one-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Female; any race or ethnicity; age 18 to 65 years old.
2. Sexual assault that occurred within the past ten weeks.
3. Subjects must be able to comprehend English.
4. Report a minimum of two substance use disorder symptoms
5. A minimum of one symptom of each cluster of Posttraumatic Stress Disorder
6. Subjects may also meet criteria for a mood disorder or other anxiety disorders (panic disorder, agoraphobia, social phobia, generalized anxiety disorder, or obsessive compulsive disorder). The inclusion of subjects with affective and other anxiety disorders is essential because of the marked frequency of the co-existence of mood and other anxiety disorders among patients with substance use disorder and posttraumatic stress disorder
7. Must consent to complete all treatment and follow-up visits.

Exclusion Criteria:

1. Lack of any memory of the sexual assault
2. Women who are menopausal
3. Subjects with a history of or current psychotic, manic, dissociative identify disorder, or a current eating disorder, as the study protocol may be therapeutically insufficient.
4. Subjects experiencing significant withdrawal symptoms, as evidence by a score of 10 or more on the Clinical Institute Withdrawal Assessment for Alcohol (CIWA)99 or a positive score of on the Clinical Opiate Withdrawal Scale.100 These subjects will be referred for clinical detoxification and may be re-assessed for study eligibility after medically supervised detoxification has been completed.
5. Individuals considered an immediate suicide risk, with current suicidal ideation and intent. These individuals will be referred directly for treatment.
6. Individuals on psychotropic medications must be stabilized on it for at least two weeks prior to beginning the study.
7. Any other medical or psychiatric conditions that the investigators believe may compromise the individual's ability to safely participate in the study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women are eligible
Enrollment: 8 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2022-08-08 (Actual); Study Completion 2022-08-08 (Actual)

PRIMARY OUTCOMES:
Change in Percent Drinking Days on The Time Line Follow-Back | Participants will report on drinking during the 30 days prior to initiation of the study, and every day until completion of study visits, approximately six weeks.
  The Time Line Follow Back (TLFB) will be used to assess heavy drinking in the past 30-days. This calendar-assisted interview yielded estimates in terms of the number of standard drinks consumed daily in the past 30 days used to obtain retrospective self-report of alcohol use by using a calendar and other memory prompts to stimulate recall.
Change in Percent Substance Use Days on The Time Line Follow-Back | Participants will report on substance use during the 30 days prior to initiation of the study, and every day until study completion of study visits, approximately six weeks.
  The Time Line Follow Back (TLFB) will be used to assess substance use in the past 30-days. This calendar-assisted interview yielded estimates in terms of the amount of substances consumed daily in the past 30 days used to obtain retrospective self-report of alcohol use by using a calendar and other memory prompts to stimulate recall.
Change in number of standard drinks per drinking day on The Time Line Follow-Back | Participants will report on drinking during the 30 days prior to initiation of the study, and ever day until completion of study visits, approximately six weeks.
  The Time Line Follow Back (TLFB) will be used to assess heavy drinking in the past 30-days and use. This calendar-assisted interview yielded estimates in terms of the number of standard drinks consumed daily in the past 30 days used to obtain retrospective self-report of alcohol use by using a calendar and other memory prompts to stimulate recall.
Change in Posttraumatic Stress Disorder Symptoms on The Posttraumatic Stress Disorder Checklist for Diagnostic Change in Posttraumatic Stress Disorder Symptoms on The Posttraumatic Stress Disorder Checklist | : Baseline and after completion of study visits, approximately six weeks.
  Participants will be asked to complete the 20-item Posttraumatic Checklist for Diagnostic and Statistical Manual of Mental Disorders (PCL-5) to measure traumatic stress symptoms corresponding with the Diagnostic and Statistical Manual of Mental Disorders -5 PTSD criteria. Items are rated on a five-point Likert scale ranging from 0 (Not at all) to 4 (Extremely) with higher scores indicating greater traumatic stress symptoms. Total scores will be used.
Change in Posttraumatic Stress Disorder Symptoms on The Clinician-Administered Posttraumatic Stress Disorder Scale for the Diagnostic and Statistical Manual of Mental Disorders | Baseline and after completion of study visits, approximately six weeks.
  The Clinician-Administered Posttraumatic Stress Disorder Scale for the Diagnostic and Statistical Manual of Mental Disorders (CAPS-5) is the gold standard in Posttraumatic Stress Disorder (PTSD) assessment. It is a structured 30-minute interview that can be used to diagnosis PTSD. Items focus on symptom presence, onset and duration of symptoms, subjective distress, impact on functioning, and symptom improvement.

SECONDARY OUTCOMES:
Change in Depression Symptoms on The Beck Depression Inventory-II | Baseline and after completion of study visits, approximately six weeks.
  The Beck Depression Inventory-II (BDI-II) is a widely used self-report measure for attitudes and symptoms of depression. The BDI-II includes 21 self-report items and takes approximately 5-minutes to complete. Each item is rated on a 4-point scale ranging from 0 to 3. The maximum total score is 63. A total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe.
Change in Anxiety Symptoms on The Beck Anxiety Inventory | Baseline and after completion of study visits, approximately six weeks.
  The Beck Anxiety Inventory (BAI) assesses symptoms of anxiety via 21-item self-report. The BAI reliability discriminates anxiety-disordered from non-anxiety disordered patients and demonstrates excellent convergence with related anxiety scales. The values for each item are summed yielding an overall or total score for all 21 symptoms that can range between 0 and 63 points. A total score of 0 - 7 is interpreted as a "Minimal" level of anxiety; 8 - 15 as "Mild"; 16 - 25 as "Moderate", and; 26 - 63 as "Severe".
Change in Depression Symptoms on The PHQ-9 | Baseline and after completion of study visits, approximately six weeks.
  The Patient Health Questionnaire (PHQ-9) is a widely used self-report measure for symptoms of depression. The PHQ-9 includes 9 self-report items, with total scores ranging from 0 to 27, and takes less than 5-minutes to complete. Scores of 5 (mild), 10 (moderate), 15 (moderately severe), and 20 (severe) are cut-off points.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No